CLINICAL TRIAL: NCT06927934
Title: Postmarketing, Prospective, Multicenter, Single-Arm Study of Subjects Who Receive an Injection of Medical Device Based on Hyaluronic Acid Marketed in Ukraine and Poland Administered Intra-Articularly to Patients Affected by Knee Osteoarthritis
Brief Title: Postmarketing Multicenter Study of Intra-Articular DIART ONE / EASYGO ONE for Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Yuria-Pharm (Industry)
Collaborators: Pharmaxi Clinical Research LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: DIART/REG-21; DIART/REG-21 (Registry Identifier: Sponsor Registry)
Record Dates: First submitted 2025-04-04; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis; Osteoarthritis of the Knee; Degenerative Joint Disease
Keywords: Hyaluronic acid; Intra-articular injection; DIART ONE; EASYGO ONE; Synovial fluid replacement; Joint pain; Single-arm study; Osteoarthritis treatment; Knee joint mobility; Degenerative joint disease; Diaco Biofarmaceutici; Yuria-Pharm
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Arthralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No samples will be retained. This study involved only clinical assessments and questionnaire-based outcomes (e.g., WOMAC index). No biological specimens were collected or stored.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study looked at how safe and effective a hyaluronic acid-based injection (called DIART ONE or EASYGO ONE) is for people with knee osteoarthritis. The injection helps replace the natural fluid in the knee joint to reduce pain and improve movement. Patients received one injection, and their symptoms were tracked over 6 months using phone calls and clinic visits. The goal was to see how much pain and joint function improved, and to check for any side effects.

DETAILED DESCRIPTION:
This was a post-marketing, observational clinical study designed to evaluate the safety, tolerability, and effectiveness of a single intra-articular injection of a stabilized hyaluronic acid-based medical device, marketed under the names DIART ONE (in Ukraine) and EASYGO ONE (in Poland). The study focused on adults diagnosed with knee osteoarthritis, a common joint disease that causes pain, stiffness, and reduced mobility due to the breakdown of joint cartilage and decreased synovial fluid.

A total of 55 participants were enrolled across multiple centers. Each participant received one injection of the investigational product into the affected knee. The specific formulation (either 20 mg/mL - 2 mL or 30 mg/mL - 3 mL) was selected by the treating physician based on clinical needs and product availability.

The primary goal of the study was to assess the change in pain levels 3 months after injection, using the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) pain subscale, a validated questionnaire used to evaluate joint pain. Secondary outcomes included changes in pain at other time points (1, 2, 4, 5, and 6 months), as well as changes in joint stiffness and physical function.

Participants were monitored over a 6-month period through a mix of in-person and phone follow-ups. Adverse events, including any side effects related to the product or injection, were documented and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years.
* Body Mass Index (BMI) ≥ 18.5 kg/m².
* Body Mass Index (BMI) < 35 kg/m².
* Presence of trauma or degenerative diseases (e.g., osteoarthritis) confirmed by radiographic imaging (Kellgren-Lawrence score 2-4).
* The subject is prescribed an injection of stabilized hyaluronic acid (DIART ONE 20 mg/mL - 2 mL or 30 mg/mL - 3 mL) for temporary replacement of synovial fluid in the knee joint.
* Signed written informed consent to participate in the study.

Exclusion Criteria:

* Age < 21 years.
* Body Mass Index (BMI) < 18.5 kg/m².
* Body Mass Index (BMI) ≥ 35 kg/m².
* Pregnancy or lactation.
* No radiographic confirmation of osteoarthritis (Kellgren-Lawrence score 0-1).
* Known hypersensitivity to hyaluronic acid, its metabolites, or excipients in the injectable implant.
* Increased bleeding tendency.
* Injury or infection at the injection site.
* Confirmed infectious joint disease.
* Systemic connective tissue diseases (e.g., active rheumatoid arthritis, ankylosing spondylitis).
* Non-osteoarthritis arthritis.
* Planned total knee joint replacement.
* Gait disorders of neurological origin.
* Intra-articular hyaluronic acid injection in the study knee within 3 months prior to enrollment.
* Surgery or orthopedic intervention on the study knee in the last 3 months.
* Cancer
* Decompensated diabetes mellitus.
* Hematological diseases.
* Inability or unwillingness to comply with study procedures.
* Language barriers that prevent understanding of the informed consent form.
* Any other condition deemed by the investigator to preclude participation.
* Participation in another clinical study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult men and women aged 21 years and older with radiographically confirmed knee osteoarthritis (Kellgren-Lawrence grade 2-4). Participants were eligible if they were prescribed a single intra-articular injection of stabilized hyaluronic acid (DIART ONE or EASYGO ONE) as part of routine clinical care for synovial fluid deficiency. All participants had a Body Mass Index (BMI) between 18.5 and 35 kg/m². Individuals with other joint diseases, recent joint surgery, infections, or contraindications to hyaluronic acid were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Change in the WOMAC Pain Subscale Score at 3 Months | 3 months after injection (Day 90 ± 5 days)
  Mean change from baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score (5-point Likert-type scale, range 0-20) at 3 months after a single intra-articular injection of hyaluronic acid.

SECONDARY OUTCOMES:
Change in the Total WOMAC Score at 1, 2, 3, 4, 5, and 6 Months | 1, 2, 3, 4, 5, and 6 months after injection
  Mean change from baseline in the total WOMAC index score (Likert-type scale, total range 0-96: pain = 0-20, stiffness = 0-8, physical functioning = 0-68) at multiple time points following injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaxi Clinical Research LLC, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No